CLINICAL TRIAL: NCT04986813
Title: Efficacy of Tranexamic Acid in Reducing Requirement of Blood Transfusion in Lower Limb Trauma Surgery: A Prospective Randomized Controlled Study
Brief Title: Tranexamic Acid in Trauma Surgery Tranexamic Acid in Trauma Surgery Tranexamic Acid in Trauma Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jaspreet Singh (Other)
Responsible Party: Sponsor-Investigator, Jaspreet Singh, Specialist Medical Officer, AP Jain Civil Hospital, Rajpura
Organization: AP Jain Civil Hospital, Rajpura (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PHMA/GSMCH-17/IEC-29A
Record Dates: First submitted 2021-07-05; First posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Tranexamic Acid; Trauma; Lower Extremity Fracture
Keywords: Tranexamic acid; Deep Vein Thrombosis; Blood transfusion
MeSH Terms: conditions — Wounds and Injuries; Venous Thrombosis | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Intervention Model Description: This was a single centre, parallel group, prospective randomized control study.
Who Masked: Participant
Masking Description: The random allocation of the patients to either group was done by one of the investigators using a random number table.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Tranexamic Acid (Active Comparator): 50 patients were given 1 gram of Tranexamic acid (TXA) intravenously pre-operatively. Intravenous TXA was administered, at the time of start of surgical incision.
  Interventions: Drug: Tranexamic acid injection
- Control group (Placebo Comparator): 50 patients were kept as a control group and were not given TXA.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: Tranexamic acid injection — 1 g of TXA in 100 ml of normal saline
  Other Names: Inj Tranexa
  Arms: Group Tranexamic Acid
Other: Normal Saline — 100 ml
  Other Names: NS
  Arms: Control group

SUMMARY:
This study was done to evaluate the efficacy of Tranexamic Acid (TXA) in reducing blood transfusion requirement in patients of lower limb trauma undergoing surgery.

DETAILED DESCRIPTION:
This was a single centre, parallel group, prospective randomized control study. 116 patients of lower limb trauma presented between April 2017 to August 2018 at Civil Hospital Rajpura. 16 patients were excluded due to old fracture, percutaneous wire fixation or non-consenting patient. The remaining 100 patients were randomized into two groups. 50 patients were given 1 gram of TXA before surgery and 50 patients were not given TXA. Fall in Hb, requirement of blood transfusion, number of days admitted in the hospital after surgery and evidence of deep vein thrombosis were monitored.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from lower limb trauma

Exclusion Criteria:

* Presence of old implant or infection at the fracture site,
* Any blood coagulation disorder
* Patients undergoing percutaneous wire placement procedures for fracture fixation
* Polytrauma
* Non-consenting patients
* Psychiatric patient

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Requirement of number of units of blood transfusion | Average of 15 days
  From the date of surgery till time of discharge

SECONDARY OUTCOMES:
Evidence of deep vein thrombosis by Wells Score | Average of 15 days (From the date of surgery till time of discharge)
  Based on Wells et al Clinical model for DVT
Change in Haemoglobin level post surgery | Average of 15 days (From the date of surgery till time of discharge)
  From the date of surgery till time of discharge
Number of days admitted in the hospital after surgery | Average of 15 days (From the date of admission till time of discharge)
  From the date of admission till time of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Gurleen Kaur, MD, Study Director — Adesh Medical College & Hospital
Locations (1):
- APJain Civil Hospital, Rajpura, Patiāla, Punjab, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaye JA, Jick H. Epidemiology of lower limb fractures in general practice in the United Kingdom. Inj Prev. 2004 Dec;10(6):368-74. doi: 10.1136/ip.2004.005843. PMID 15583259
- [Result] Zhang P, Bai J, He J, Liang Y, Chen P, Wang J. A systematic review of tranexamic acid usage in patients undergoing femoral fracture surgery. Clin Interv Aging. 2018 Sep 4;13:1579-1591. doi: 10.2147/CIA.S163950. eCollection 2018. PMID 30233155
- [Result] Fischer PE, Bulger EM, Perina DG, Delbridge TR, Gestring ML, Fallat ME, Shatz DV, Doucet J, Levy M, Stuke L, Zietlow SP, Goodloe JM, VanderKolk WE, Fox AD, Sanddal ND. Guidance Document for the Prehospital Use of Tranexamic Acid in Injured Patients. Prehosp Emerg Care. 2016 Sep-Oct;20(5):557-9. doi: 10.3109/10903127.2016.1142628. Epub 2016 Mar 17. PMID 26985786

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-05): https://cdn.clinicaltrials.gov/large-docs/13/NCT04986813/Prot_SAP_000.pdf